CLINICAL TRIAL: NCT04254094
Title: Study of Behavioural and Psychological Symptoms as Functional Prognostic Factors in Neurodegenerative Early Onset Major Neurocognitive Disorders
Brief Title: A Cohort Study of Early Onset Neurodegenerative Dementias Prognostic Factors
Acronym: NEODEM
Status: Active, not recruiting | Type: Observational
Sponsor: University Hospital, Bordeaux (Other)
Responsible Party: Sponsor
Other Study IDs: CHUBX 2018/68
Record Dates: First submitted 2020-01-31; First posted 2020-02-05 (Actual); Last update posted 2023-10-06 (Actual); Status verified 2023-10

CONDITIONS: Dementia
MeSH Terms: conditions — Dementia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 36 Months
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Early onset dementias (EOD): Prospective multicenter cohort of EOD patients with a three-year follow-up in tertiary Reference Memory centers
  Interventions: Other: Neuropsychological scales

INTERVENTIONS:
Other: Neuropsychological scales — Basic Activity of Daily Living (BADL) and Instrumental Activities of Daily Living (IADL), Neuropsychiatric Inventory (NPI), Cornell Scale for Depression in Dementia (CSDD), Clinical Dementia Rating Scale (CDR) and defining dementia criteria. Also as part of this study, an MRI examination at baseline and at 18 months follow-up will be performed in the Bordeaux center

SUMMARY:
NEODEM is a multicenter cohort study of patients with early-onset degenerative dementia (before age 65), the main objective of which is to study behavioral disorders and in particular depression as functional prognostic factors at 3 years.

DETAILED DESCRIPTION:
Early-onset dementia (EOD), which begins before the age of 65, is less common than late-onset dementia but represents a significant burden for the patient, their family and the healthcare system. The descriptive epidemiology is poorly known, and the National Reference Center for young patients, using English data (Harvey et al., 2003) estimates the number of subjects concerned in France at 18,318. It is degenerative dementia that is the most common cause of EOD and among them, Alzheimer's disease and then frontotemporal degeneration (FTD) (Vieira et al., 2013). The natural history and prognostic factors of PDD are not well known, and only AD has some data. Alzheimer's disease (AD) in young people appears to have a worse prognosis than that in older people, but this is debated (Stanley and Walker, 2014) and also depends on the criteria studied: cognition, function or survival. Prognostic factors other EOD, and in particular frontotemporal dementias, which moreover are heterogeneous pathologies, are even less known.

Investigators have chosen to study the functional prognosis of patients because it is both very relevant to care needs and easy to measure. Among the prognostic factors of functional status, investigators will study in particular psycho-behavioral disorders, and in particular depression, which is very common in patients with EOD, a factor of poor quality of life and accessible to treatment. Other potential prognostic factors such as cognitive reserve, gender, clinical variants of AD and DFT, family status (living alone or having a caregiver), genetic status, family history of dementia, CSF biomarkers and MRI imaging will be studied . The evolution of instrumental activities of daily living will be measured. The social and paramedical resources used by the patient and his family will be collected, as well as the use of psychotropic and non-drug treatments. Finally, the overall evolution of the severity of dementia will be measured.

Eligible patients will be included for 3 years and evaluated every 6 months.

ELIGIBILITY:
Inclusion Criteria:

1. Newly diagnosed neurodegenerative (within 6 months) EOD according to international consensus criteria
2. Symptoms onset before 65 years old
3. Clinical Dementia Rating Scale (CDR) 0.5 to 1 both inclusive
4. Affiliated person or beneficiary of a social security scheme.
5. Free and informed consent obtained and signed by the patient or by the patient's representative and a non-opposition letter signed by the caregiver when available
6. Able to participate to cognitive and psychiatric assessments

Exclusion Criteria:

1. Non degenerative dementias : e;g. vascular, alcohol-related, toxic, infectious, posttraumatic.
2. Dementia of unknown etiology
3. Dementia in Down syndrome
4. Patients in Nursing Home or other care facility
5. Total dependency for dressing and/or bathing at the time of inclusion
6. Patient with a severe or life-threatening disease

   -

Ages: 18 Years to 65 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Newly diagnosed neurodegenerative (within 6 months) EOD according to international consensus criteria with symptoms onset before 65 years old
Sampling Method: Non-Probability Sample
Enrollment: 163 (Actual)
Dates: Start 2020-05-20 (Actual); Primary Completion 2026-05-20 (Estimated); Study Completion 2026-05-20 (Estimated)

PRIMARY OUTCOMES:
BADL dependency in both bathing and dressing using the BADL scale from Katz (Katz et al., 1970) at inclusion | at inclusion
  Katz scale ranks the adequacy of performance in six basic functions including bathing, dressing, toileting, transferring,continence, and feeding.. It has been shown that bathing and dressing are the first ADL to be lost, also defined by Katz et al. as the thresholds for disability (Katz et al., 1970 ; Edjolo et al., 2016). Each item is graded according to the level of dependence as follows: performs independently (0 point), performs with assistance (1 point), and unable to perform (2 point). A total score of 0 indicates "full function" and 12 indicates "severe functional impairment". To evaluate the primary outcome, only the score at the two first items (bathing and dressing, scoring from 0 to 4) will be taken into account for the analysis: complete dependency is present if the score at the two first items is 4 and absent if <4.
BADL dependency in both bathing and dressing using the BADL scale from Katz (Katz et al., 1970) at 6 months | 6 months after inclusion
  Katz scale ranks the adequacy of performance in six basic functions including bathing, dressing, toileting, transferring,continence, and feeding.. It has been shown that bathing and dressing are the first ADL to be lost, also defined by Katz et al. as the thresholds for disability (Katz et al., 1970 ; Edjolo et al., 2016). Each item is graded according to the level of dependence as follows: performs independently (0 point), performs with assistance (1 point), and unable to perform (2 point). A total score of 0 indicates "full function" and 12 indicates "severe functional impairment". To evaluate the primary outcome, only the score at the two first items (bathing and dressing, scoring from 0 to 4) will be taken into account for the analysis: complete dependency is present if the score at the two first items is 4 and absent if <4.
BADL dependency in both bathing and dressing at 12 months | 12 months after inclusion
  Katz scale ranks the adequacy of performance in six basic functions including bathing, dressing, toileting, transferring,continence, and feeding.. It has been shown that bathing and dressing are the first ADL to be lost, also defined by Katz et al. as the thresholds for disability (Katz et al., 1970 ; Edjolo et al., 2016). Each item is graded according to the level of dependence as follows: performs independently (0 point), performs with assistance (1 point), and unable to perform (2 point). A total score of 0 indicates "full function" and 12 indicates "severe functional impairment". To evaluate the primary outcome, only the score at the two first items (bathing and dressing, scoring from 0 to 4) will be taken into account for the analysis: complete dependency is present if the score at the two first items is 4 and absent if <4.
BADL dependency in both bathing and dressing at 18 months | 18 months after inclusion
  Katz scale ranks the adequacy of performance in six basic functions including bathing, dressing, toileting, transferring,continence, and feeding.. It has been shown that bathing and dressing are the first ADL to be lost, also defined by Katz et al. as the thresholds for disability (Katz et al., 1970 ; Edjolo et al., 2016). Each item is graded according to the level of dependence as follows: performs independently (0 point), performs with assistance (1 point), and unable to perform (2 point). A total score of 0 indicates "full function" and 12 indicates "severe functional impairment". To evaluate the primary outcome, only the score at the two first items (bathing and dressing, scoring from 0 to 4) will be taken into account for the analysis: complete dependency is present if the score at the two first items is 4 and absent if <4.
BADL dependency in both bathing and dressing at 24 months | 24 months after inclusion
  Katz scale ranks the adequacy of performance in six basic functions including bathing, dressing, toileting, transferring,continence, and feeding.. It has been shown that bathing and dressing are the first ADL to be lost, also defined by Katz et al. as the thresholds for disability (Katz et al., 1970 ; Edjolo et al., 2016). Each item is graded according to the level of dependence as follows: performs independently (0 point), performs with assistance (1 point), and unable to perform (2 point). A total score of 0 indicates "full function" and 12 indicates "severe functional impairment". To evaluate the primary outcome, only the score at the two first items (bathing and dressing, scoring from 0 to 4) will be taken into account for the analysis: complete dependency is present if the score at the two first items is 4 and absent if <4.
BADL dependency in both bathing and dressing at 30 months | 30 months after inclusion
  Katz scale ranks the adequacy of performance in six basic functions including bathing, dressing, toileting, transferring,continence, and feeding.. It has been shown that bathing and dressing are the first ADL to be lost, also defined by Katz et al. as the thresholds for disability (Katz et al., 1970 ; Edjolo et al., 2016). Each item is graded according to the level of dependence as follows: performs independently (0 point), performs with assistance (1 point), and unable to perform (2 point). A total score of 0 indicates "full function" and 12 indicates "severe functional impairment". To evaluate the primary outcome, only the score at the two first items (bathing and dressing, scoring from 0 to 4) will be taken into account for the analysis: complete dependency is present if the score at the two first items is 4 and absent if <4.
BADL dependency in both bathing and dressing at 36 months | 36 months after inclusion
  Katz scale ranks the adequacy of performance in six basic functions including bathing, dressing, toileting, transferring,continence, and feeding.. It has been shown that bathing and dressing are the first ADL to be lost, also defined by Katz et al. as the thresholds for disability (Katz et al., 1970 ; Edjolo et al., 2016). Each item is graded according to the level of dependence as follows: performs independently (0 point), performs with assistance (1 point), and unable to perform (2 point). A total score of 0 indicates "full function" and 12 indicates "severe functional impairment". To evaluate the primary outcome, only the score at the two first items (bathing and dressing, scoring from 0 to 4) will be taken into account for the analysis: complete dependency is present if the score at the two first items is 4 and absent if <4.

SECONDARY OUTCOMES:
Behavioral and Psychological Symptoms of Dementia (BPSD) as measured by Neuropsychiatric Inventory (NPI) at the inclusion | at the inclusion
  The NPI is a caregiver administered scale which assesses 12 domains of BPSD in dementia (Cummings et al., 1994). The NPI has been validated in French (Robert et al., 1998) . It is a questionnaire composed of a screening question and seven to nine items for each of 12 domains : delusions, hallucinations, agitation/aggression, depression/dysphoria, anxiety, elation/euphoria, apathy/indifference, disinhibition, irritability/lability, aberrant motor behavior, sleep, appetite and eating disorders. A knowledgeable informant (usually a caregiver) indicates via the screening question whether the patient has experienced any domain-related symptom in the past month. If the screening question is validated, the caregiver is then asked whether each item within the domain has occurred in the past month and provides a global rating of frequency, severity and caregiver distress for all items in the domain at the same time (not item by item). Score ranges from 0 to 144 .
BPSD as measured by NPI at 12 months after inclusion | at 12 months after inclusion
  The NPI is a caregiver administered scale which assesses 12 domains of BPSD in dementia (Cummings et al., 1994). The NPI has been validated in French (Robert et al., 1998) . It is a questionnaire composed of a screening question and seven to nine items for each of 12 domains : delusions, hallucinations, agitation/aggression, depression/dysphoria, anxiety, elation/euphoria, apathy/indifference, disinhibition, irritability/lability, aberrant motor behavior, sleep, appetite and eating disorders. A knowledgeable informant (usually a caregiver) indicates via the screening question whether the patient has experienced any domain-related symptom in the past month. If the screening question is validated, the caregiver is then asked whether each item within the domain has occurred in the past month and provides a global rating of frequency, severity and caregiver distress for all items in the domain at the same time (not item by item). Score ranges from 0 to 144 .
BPSD as measured by NPI at 24 months after inclusion | at 24 months after inclusion
  The NPI is a caregiver administered scale which assesses 12 domains of BPSD in dementia (Cummings et al., 1994). The NPI has been validated in French (Robert et al., 1998) . It is a questionnaire composed of a screening question and seven to nine items for each of 12 domains : delusions, hallucinations, agitation/aggression, depression/dysphoria, anxiety, elation/euphoria, apathy/indifference, disinhibition, irritability/lability, aberrant motor behavior, sleep, appetite and eating disorders. A knowledgeable informant (usually a caregiver) indicates via the screening question whether the patient has experienced any domain-related symptom in the past month. If the screening question is validated, the caregiver is then asked whether each item within the domain has occurred in the past month and provides a global rating of frequency, severity and caregiver distress for all items in the domain at the same time (not item by item). Score ranges from 0 to 144 .
BPSD as measured by NPI at 36 months after inclusion | at 36 months after inclusion
  The NPI is a caregiver administered scale which assesses 12 domains of BPSD in dementia (Cummings et al., 1994). The NPI has been validated in French (Robert et al., 1998) . It is a questionnaire composed of a screening question and seven to nine items for each of 12 domains : delusions, hallucinations, agitation/aggression, depression/dysphoria, anxiety, elation/euphoria, apathy/indifference, disinhibition, irritability/lability, aberrant motor behavior, sleep, appetite and eating disorders. A knowledgeable informant (usually a caregiver) indicates via the screening question whether the patient has experienced any domain-related symptom in the past month. If the screening question is validated, the caregiver is then asked whether each item within the domain has occurred in the past month and provides a global rating of frequency, severity and caregiver distress for all items in the domain at the same time (not item by item). Score ranges from 0 to 144 .
Depression as measured by the Cornell Scale for Depression in Dementia at inclusion | at inclusion
  the Cornell Scale for Depression in Dementia is a 19-item clinician-administered instrument that uses information from interviews with both the patient and an informant, specifically designed for the rating of symptoms of depression in demented patients (Alexopoulos et al., 1988). Items were constructed so they can be rated primarily on the basis of observation, and not self report by the patient. The severity of each item is described as absent, mild or intermittent, and severe. The informant is interviewed first. Time of administration is about 30 minutes. The CSDD has been validated in French (Camus et al., 1995). Mean scores are given in the original paper, as a function of MMSE for no depression, episodic minor depressive disorder, probable major depressive disorder and definite major depressive disorder.
Depression as measured by the Cornell Scale for Depression in Dementia at 12 months after inclusion | at 12 months after inclusion
  the Cornell Scale for Depression in Dementia is a 19-item clinician-administered instrument that uses information from interviews with both the patient and an informant, specifically designed for the rating of symptoms of depression in demented patients (Alexopoulos et al., 1988). Items were constructed so they can be rated primarily on the basis of observation, and not self report by the patient. The severity of each item is described as absent, mild or intermittent, and severe. The informant is interviewed first. Time of administration is about 30 minutes. The CSDD has been validated in French (Camus et al., 1995). Mean scores are given in the original paper, as a function of MMSE for no depression, episodic minor depressive disorder, probable major depressive disorder and definite major depressive disorder.
Depression as measured by the Cornell Scale for Depression in Dementia at 24 months after inclusion | at 24 months after inclusion
  the Cornell Scale for Depression in Dementia is a 19-item clinician-administered instrument that uses information from interviews with both the patient and an informant, specifically designed for the rating of symptoms of depression in demented patients (Alexopoulos et al., 1988). Items were constructed so they can be rated primarily on the basis of observation, and not self report by the patient. The severity of each item is described as absent, mild or intermittent, and severe. The informant is interviewed first. Time of administration is about 30 minutes. The CSDD has been validated in French (Camus et al., 1995). Mean scores are given in the original paper, as a function of MMSE for no depression, episodic minor depressive disorder, probable major depressive disorder and definite major depressive disorder.
Depression as measured by the Cornell Scale for Depression in Dementia at 36 months after inclusion | at 36 months after inclusion
  the Cornell Scale for Depression in Dementia is a 19-item clinician-administered instrument that uses information from interviews with both the patient and an informant, specifically designed for the rating of symptoms of depression in demented patients (Alexopoulos et al., 1988). Items were constructed so they can be rated primarily on the basis of observation, and not self report by the patient. The severity of each item is described as absent, mild or intermittent, and severe. The informant is interviewed first. Time of administration is about 30 minutes. The CSDD has been validated in French (Camus et al., 1995). Mean scores are given in the original paper, as a function of MMSE for no depression, episodic minor depressive disorder, probable major depressive disorder and definite major depressive disorder.
Institutionalization | at 36 months after inclusion
  date of institutionalization
Death | at 36 months after inclusion
  date of death
BPSD other than depression at inclusion | at inclusion
  Neuropsychiatric Inventory with an informant if any (de Medeiros et al., 2010). This scale will be administered by an experienced clinician or psychologist. Both the subscore of each of the 12 domains and the total score will be analysed
BPSD other than depression at 12 months after inclusion | at 12 months after inclusion
  Neuropsychiatric Inventory with an informant if any (de Medeiros et al., 2010). This scale will be administered by an experienced clinician or psychologist. Both the subscore of each of the 12 domains and the total score will be analysed
BPSD other than depression at 24 months after inclusion | at 24 months after inclusion
  Neuropsychiatric Inventory with an informant if any (de Medeiros et al., 2010). This scale will be administered by an experienced clinician or psychologist. Both the subscore of each of the 12 domains and the total score will be analysed
BPSD other than depression at 36 months after inclusion | at 36 months after inclusion
  Neuropsychiatric Inventory with an informant if any (de Medeiros et al., 2010). This scale will be administered by an experienced clinician or psychologist. Both the subscore of each of the 12 domains and the total score will be analysed

CONTACTS AND LOCATIONS:
Overall Officials: Sophie AURIACOMBE, M.D, Principal Investigator — University Hospital, Bordeaux
Locations (1):
- CHU de Bordeaux, Bordeaux, France

IPD SHARING:
Plan to Share IPD: No